CLINICAL TRIAL: NCT05387525
Title: A Phase 4, Multi-centre, Randomized, Evaluator-blinded, Active-controlled Study to Determine the Incidence of Squamous Cell Carcinoma and Evaluate the Long-term Safety of Tirbanibulin 10 mg/g Ointment and Diclofenac Sodium 3% Gel for the Treatment of Adult Patients With Actinic Keratosis on the Face or Scalp
Brief Title: A Study of Tirbanibulin Ointment and Diclofenac Sodium Gel for the Treatment of Adult Participants With Actinic Keratosis on the Face or Scalp
Acronym: AKtive
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-14789-41; 2021-004349-18 (EudraCT Number)
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic | interventions — tirbanibulin; Ointments; Diclofenac; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirbanibulin 10 milligram per gram (mg/g) ointment (Experimental): Participants will apply tirbanibulin ointment 10 mg/g once daily to the treatment field (TF) for 5 consecutive days beginning Day 1. At subsequent visits, participants will have the option of an additional 5-day course(s) (with at least 16 weeks between starting date of treatment courses) at the discretion of the investigator if actinic keratosis (AK) lesions are present in the TF and physical treatment is not appropriate.
  Interventions: Drug: Tirbanibulin (Klisyri®) 10 mg/g ointment
- Diclofenac Sodium 3% Gel (Active Comparator): Participants will apply diclofenac sodium 3% gel twice daily to the TF for 60 to 90 days beginning Day 1, with the option of further courses every 6 months (with at least 6 months between starting date of treatment courses) if lesions are found to be present in the TF at follow up visits and physical treatment is not appropriate.
  Interventions: Drug: Diclofenac Sodium 3% Gel

INTERVENTIONS:
Drug: Tirbanibulin (Klisyri®) 10 mg/g ointment — Participants will apply tirbanibulin 10 mg/g ointment topically for 5 days over 25 cm^2 of the face or scalp with Actinic Keratosis (AK).
  Other Names: Klisyri®
  Arms: Tirbanibulin 10 milligram per gram (mg/g) ointment
Drug: Diclofenac Sodium 3% Gel — Participants will apply diclofenac dodium 3% gel twice daily for 60 to 90 days.
  Arms: Diclofenac Sodium 3% Gel

SUMMARY:
The purpose of the study is to evaluate the incidence of biopsy confirmed invasive squamous cell carcinoma (SCC) in the selected treatment field (TF) after administration of topical tirbanibulin 10 milligram (mg)/gram (g) ointment or diclofenac sodium 3 percent (%) gel over the 3-year study period.

ELIGIBILITY:
Inclusion Criteria:

* A treatment field (TF) on the face or scalp (excluding lips, eyelids, ears, and inside the nostrils), that: a) is a contiguous area measuring 25 cm^2, b) contains 2 to 8 clinically typical, visible, and discrete actinic keratosis (AK) lesions, and c) has an overall clinical picture that is consistent with Olsen grade 1
* If a women of child-bearing potential (WOCBP), that is, fertile, defined as a female in the life period from menarche and until becoming post-menopausal (no menses for 12 months without an alternative medical cause) or permanently sterile (with hysterectomy, bilateral salpingectomy or bilateral oophorectomy at least 3 months prior to Screening), she must: a) Have a negative urine pregnancy test using a highly sensitive method at screening and on Day 1 prior to treatment administration. b) Be using effective methods of birth control. c) Agree to have pregnancy tests while in the study and at the end of the study
* Participants should be willing to avoid sunlight or ultraviolet (UV) light exposure, including the use of tanning beds, to the face or scalp during the study
* Participants should have the ability to understand the purpose and risks of the study, willingness and ability to comply with the protocol, and provide written informed consent in accordance with institutional and regulatory guidelines

Exclusion Criteria:

* The location of the TF is: a) on any location other than the face or scalp. b) within 5 centimeters (cm) of an incompletely healed wound. c) Within 10 cm of a suspected basal cell carcinoma (BCC) or other neoplasm. d) on the lips, eyelids, ears, or inside the nostrils, periorbital, perioral, or the skin surrounding the nostrils
* Presence in the TF of: a) clinically atypical and/or rapidly changing AK lesions b) hyperkeratotic or hypertrophic lesions, recalcitrant disease (had cryosurgery on 2 previous occasions), and/or cutaneous horn. c) confluent AK lesions (that is, non-discrete lesions, as per inclusion criterion 2). d) Persisting AK lesions at the screening visit following topical treatment with diclofenac sodium 3 percent (%) gel
* History of any malignant skin tumour in the TF or history of skin tumour in any region of the body which has metastasized or in which metastasis within the study period is likely
* History of any malignant tumour with systemic antitumor treatment (including radiotherapy) within 12 weeks prior to the Screening Visit or systemic antitumor treatment is expected while on the study
* Immunocompromised participants, including participants with a history of chronic systemic lymphoma or chronic myeloid leukaemia, or organ transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Histologically Confirmed Invasive Squamous Cell Carcinoma (SCC) in the Treatment Field (TF) | Up to 3 years
  Percentage of participants with histologically confirmed invasive SCC in the TF will be reported as assessed by dermoscopy.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 3 years
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered an Investigational Product. An AE does not necessarily have a causal relationship with the medicinal product.
Number of Participants With Serious Adverse Events (SAEs) | Up to 3 years
  A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that at any dose, resulted in death, was life-threatening (i.e, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Percentage of Participants With any Other Skin Cancer (Other Than SCC) in the TF | Up to 3 years
  Percentage of participants with any other skin cancer (other than SCC) in the TF will be reported.
Time to Occurrence of Invasive SCC From Baseline in the TF | Up to 3 years
  Time to occurrence of invasive SCC from baseline in the TF will be reported.
Percentage of Participants Requiring Rescue Treatment After 1 Treatment Course | Up to 3 years
  Percentage of participants requiring rescue treatment after 1 treatment course will be reported.
Percentage of Participants Requiring Rescue Treatment at Any Time During the Study | Up to 3 years
  Percentage of participants requiring rescue treatment at any time during the study will be reported.
Percentage of Participants With no Lesions After Treatment of the First Recurrence With Tirbanibulin During the First 52 Weeks | Up to Week 52
  Percentage of participants with no lesions after treatment of the first recurrence with tirbanibulin during the first 52 weeks will be reported.
Number of Participants With Vital Signs Abnormalities | Up to 3 years
  Number of participants with vital signs (including measurement of heart rate, respiratory rate, systolic and diastolic blood pressure and tympanic temperature) will be reported.
Number of Participants With Physical Examination Abnormalities | Up to 3 years
  Number of participants with physical examination abnormalities (height, weight and an assessment of head, eyes, ears, nose and throat, integumentary/dermatological, gastrointestinal, cardiovascular, respiratory, musculoskeletal, and neurological systems) will be reported.

CONTACTS AND LOCATIONS:
Locations (49):
- France (6):
  - Almirall Investigation Site 102, Lille
  - Almirall Investigation Site 103, Marseille
  - Almirall Investigation Site 104, Nice
  - Almirall Investigational Site 106, Paris
  - Almirall Investigational Site 105, Rouen
  - Almirall Investigational Site 101, Saint-Priest-en-Jarez
- Germany (13):
  - Almirall Investigational Site 205, Augsburg
  - Almirall Investigational Site 211, Bad Bentheim
  - Almirall Investigation Site 201, Bochum
  - Almirall Investigational Site 214, Bochum
  - Almirall Investigational Site 212, Bonn
  - Almirall Investigational Site 208, Detmold
  - Almirall Investigational Site 210, Dresden
  - Almirall Investigational Site 204, Erlangen
  - Almirall Investigational Site 206, Hamburg
  - Almirall Investigational Site 213, Hamburg
  - Almirall Investigational Site 207, Marburg
  - Almirall Investigational Site 209, Merzig
  - Almirall Investigation Site 202, Recklinghausen
- Italy (10):
  - Almirall Investigational Site 309, Arezzo
  - Almirall Investigational Site 302, Brescia
  - Almirall Investigational Site 304, Genova
  - Almirall Investigational Site 308, Modena
  - Almirall Investigational Site 301, Napoli
  - Almirall Investigational Site 303, Reggio Emilia
  - Almirall Investigational Site 305, Roma
  - Almirall Investigational Site 306, Roma
  - Almirall Investigational Site 307, Roma
  - Almirall Investigational Site 310, Rozzano
- Poland (5):
  - Almirall Investigational Site 403, Lublin
  - Almirall Investigational Site 406, Rzeszów
  - Almirall Investigational Site 407, Warsaw
  - Almirall Investigational Site 401, Wroclaw
  - Almirall Investigational Site 402, Wroclaw
- Spain (10):
  - Almirall Investigational Site 502, Barcelona
  - Almirall Investigational Site 508, Barcelona
  - Almirall Investigational Site 510, Barcelona
  - Almirall Investigational Site 507, Granada
  - Almirall Investigational Site 509, Granada
  - Almirall Investigational Site 503, Madrid
  - Almirall Investigational Site 504, Salamanca
  - Almirall Investigational Site 505, Seville
  - Almirall Investigational Site 506, Valencia
  - Almirall Investigational Site 501, Zaragoza
- United Kingdom (5):
  - Almirall Investigational Site 703, London
  - Almirall Investigational Site 709, London
  - Almirall Investigational Site 708, Oxford
  - Almirall Investigational Site 704, Poole
  - Almirall Investigational Site 706, Weston-super-Mare

IPD SHARING:
Plan to Share IPD: No